CLINICAL TRIAL: NCT00459316
Title: Phase I/II Study of Safety and Immunogenicity of Quadrivalent Meningococcal Conjugate Vaccine (MCV4) in HIV-Infected Children and Youth And Open Label Immunogenicity Study of a Booster Dose of MCV4 in Previously Immunized HIV-Infected Children and Youth
Brief Title: Safety of and Immune Response to a Meningitis Vaccine in HIV-Infected Children and Youth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P1065; 10396 (Registry Identifier: DAIDS ES Registry Number); IMPAACT P1065; PACTG P1065
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Meningitis
MeSH Terms: conditions — HIV Infections; Meningitis

ARMS (3):
- Group 1 (Experimental): Participants ≤11 to <25 years of age with CD4% at screening ≥15%. All received Quadrivalent meningococcal conjugate vaccine at entry, those who were eligible were randomized at week 24, with Group 1B receiving a second Quadrivalent meningococcal conjugate vaccine at week 24. Those who were eligible received a booster dose of Quadrivalent meningococcal vaccine at 3.5 years.
  Interventions: Biological: Quadrivalent meningococcal conjugate vaccine
- Group 2 (Experimental): Participants ≤11 to <25 years of age with CD4% at screening <15%; All receiving Quadrivalent meningococcal conjugate vaccine at entry, with those who were eligible receiving Quadrivalent meningococcal conjugate vaccine at week 24 and 3 years.
  Interventions: Biological: Quadrivalent meningococcal conjugate vaccine
- Group 3 (Experimental): Participants >=2 to <11 years of age with CD4% at screening ≥ 25%; All received Quadrivalent meningococcal conjugate vaccine at entry, with those who were eligible receiving Quadrivalent meningococcal conjugate vaccine at week 24 and 3 years.
  Interventions: Biological: Quadrivalent meningococcal conjugate vaccine

INTERVENTIONS:
Biological: Quadrivalent meningococcal conjugate vaccine — MCV4 vaccine (4 µg each of meningococcal A, C, Y, and W-135 polysaccharides conjugated to approximately 48 µg of diphtheria toxoid protein carrier ) was given by injection intramuscularly at least once and no more than three times for each participant, depending on adverse reactions.
  Other Names: MCV4

SUMMARY:
Bacterial meningitis infection is common in youth 2 to 24 years of age in the United States. This disease can be treated by antibiotics, but mortality rates associated with meningitis of up to 53% have been estimated. Vaccination against meningitis may be effective in preventing this disease, especially for HIV-infected youth who have weakened immune systems. The purpose of this study was to determine the safety of and immune response to a preventive meningitis vaccine in HIV-infected youth.

DETAILED DESCRIPTION:
In the United States, youth 2 to 24 years of age are at high risk for bacterial meningitis infection. Despite antibiotic treatment, the mortality rate for meningitis and sepsis can reach as high as 53% caused by Neisseria meningitidis. This rate could be higher in immunocompromised individuals, such as those infected with HIV. To prevent infection, vaccination against meningitis is recommended by the CDC at ages 11, 15, and 18. The quadrivalent meningococcal conjugate vaccine (MCV4) is a vaccine that has been observed to elicit an appropriate immune response to N. meningitidis and was approved by the FDA in January 2005. However, to date, no studies have been done to determine the safety and immunogenicity of this vaccine in HIV-infected individuals. The purpose of this study was to determine the safety and immunogenicity of MCV4 in HIV-infected youth 2 to 24 years of age.

The study was originally designed for participants to be followed for 72 weeks. Participants were enrolled in three groups by age and CD4% as follows:

Group 1: Age 11 to 24 years, CD4% of 15% or higher. Enrollment was further stratified by CD4%: 15% to <25%, and >= 25%.

Group 2: Age 11 to 24 years, CD4% < 15%.

Group 3: Age 2 to 10 years, CD4% of 25% or higher.

At study entry, all study participants received one injection of MCV4 (Step 1). Participants were observed for 30 minutes post-injection to monitor for adverse events. A clinic visit was required 24 hours post-injection if the participant reported adverse events. At Week 24, participants in Group 1 who did not experience any disqualifying adverse events after the first injection were randomly assigned to receive a second injection of MCV4 or no further injections. Group 2, and Group 3 participants who had no disqualifying adverse events after the first injection received a second injection of MCV4 at Week 24 (Step 2).

There were five study visits in Steps 1 and 2; they occurred at study entry and at Weeks 4, 24, 28, and 72. At these visits, a physical exam, assessment of HIV-related symptoms, and blood collection occurred. In addition, study participants were contacted by telephone at Days 3 and 7 and Weeks 1, 6, and 25 after the first vaccination. Participants in Groups 1B and 2 who received a second injection were contacted by telephone at Weeks 30 and 48.

As of November 2010, due to data from this study (P1065) and recommendations from the Advisory Committee for Immunization Practices (ACIP) of the Center for Disease Control (CDC), eligible participants in Groups 1 (1A and 1B) and 3 of P1065 received a booster dose of MCV4 at approximately 3.5 years (+/- 6 months) after the initial MCV4 vaccination. Participants were then observed for 30 minutes post-injection to monitor for adverse events. Participants were also observed at Week 1 for vaccine adverse reactions.

This portion of the study (Step 3) lasted an additional 24 weeks. There were 4 study visits; they occurred at entry, at Days 7-8, and at Weeks 4 and 24. At these visits, a physical exam, assessment of HIV-related symptoms, and blood collection occurred. The purpose of this follow-up study was to determine the safety and immunogenicity of a MCV4 booster dose in HIV-infected participants who have previously received one or two MCV4 vaccinations on this study.

ELIGIBILITY:
Inclusion Criteria for Steps 1, 2, and 3:

* HIV-infected
* Age greater than or equal to 2 and less than 25 years (Steps 1 and 2 only)
* CD4% documented within 120 days of study entry
* Participants on antiretroviral therapy (ART) must have been on stable ART regimen for at least 90 days prior to study entry
* Able and willing to complete all study immunizations and evaluations
* Parent or guardian willing to provide informed consent, if applicable
* Participants and/or their partners who are sexually active had to agree to use at least one of the following methods of contraception as long as they are on the study: hormonal birth control drugs (oral, injectable or transdermal); male or female condoms with or without a spermicide; diaphragm/cervical cap with spermicide; intrauterine device (IUD)

Inclusion Criteria specific to Step 3:

* Participants must have been enrolled in Groups 1 or 3 of previous versions of P1065
* Participants did not have to be less than 25 years of age
* Participants must have had serology data from Weeks 0, 4, and 28 from their previous participation in P1065
* Participants must have been within 3.5 years +/- 6 months from the first MCV4 dose received in a previous version of P1065

Exclusion Criteria for Step 1:

* Any nonstudy vaccine on study entry day
* Any inactive vaccine within 2 weeks prior to study entry
* Plans to receive any vaccine 2 weeks after the first injection
* Receipt of any live nonstudy vaccine within 4 weeks prior to study entry
* Meningococcal conjugate vaccine at any time prior to study entry
* Meningococcal polysaccharide vaccine within 2 years prior to study entry
* Known hypersensitivity to any component of the MCV4 vaccine, including diphtheria toxoid
* Known hypersensitivity to dry natural rubber latex
* Life-threatening reaction after previous administration of a vaccine containing similar components
* Family history or personal history of Guillain-Barre Syndrome (GBS)
* Clinically significant diseases that, in the investigator's opinion, would interfere with the study
* Current immunomodulatory therapy, including IL-2, any interferon product, GM-CSF, or thalidomide. Participants taking G-CSF or erythropoietin were not excluded.
* Current immunosuppressive therapy, including equivalent of 1 mg/kg/per day or more of prednisone 2 weeks prior to study entry OR planned corticosteroid therapy lasting 2 weeks or longer. Participants using nonsteroidal anti-inflammatory agents and inhaled corticosteroids are not excluded.
* Cancer within 12 weeks of study entry
* Cancer treatment currently or within 12 weeks of study entry
* Loss of strength in lower extremity within 24 weeks prior to study entry
* Bleeding disorder or anticoagulant therapy prior to study entry
* Absence of ankle and patellar deep tendon reflexes (DTRs) (all four)
* Recent receipt of IGIV or any blood or immunoglobulin product (except washed blood cells). More information about this criterion can be found in the protocol.
* Other acute or chronic medical or surgical conditions or contraindications that, in the opinion of the investigator, might have interfered with the study
* Any new and unresolved Grade 3 or higher laboratory toxicity within 120 days prior to study entry
* Any new and unresolved Grade 3 or higher clinical toxicity within 120 days prior to study entry
* Pregnancy or breastfeeding

Exclusion Criteria for Step 2:

* New occurrence or awareness of GBS in the participant or participant's family since study entry
* Loss of strength in lower extremity or extremities since first vaccination
* Absence of ankle and patellar DTRs (all four)
* New diagnosis of active cancer, or chemotherapy treatment of an established cancer diagnosis since study entry
* Any Grade 4 toxicity since last vaccination. Participants who experience toxicities unrelated to the vaccine are not excluded.
* Change in ART in the 90 days prior to second vaccination
* Certain Grade 3 toxicities. More information on this criterion can be found in the protocol.
* Treatment with immunosuppressive or immunomodulation therapy (other than corticosteroids) within 60 days of planned second vaccination
* Severe allergic reaction requiring medical intervention within 24 hours of the first vaccination
* New diagnosis of any coagulation disorder that would contraindicate intramuscular injection
* Toxicity from first vaccination. More information on this criterion can be found in the protocol.
* Any new diseases that the investigator judges to be clinically significant OR clinically significant findings since the first vaccination that, in the opinion of the investigator, would interfere with the study
* Any new clinical Grade 3 or higher toxicity that has not resolved within 2 weeks prior to planned second vaccination
* Pregnancy or breastfeeding. Pregnant or breastfeeding participants were to be followed to pregnancy outcome.

Exclusion Criteria for Step 3:

* Receipt of any dose of non-study meningococcal vaccine since initial enrollment into P1065
* New occurrence or new awareness of GBS in the participant or participant's family since the last P1065 study visit
* Loss of strength in lower extremity or extremities since the last MCV4 vaccination
* Absence of ankle and patellar Deep Tendon Reflexes (DTRs) (all 4)
* New diagnosis of an active malignancy, or chemotherapy treatment of an established diagnosis since the last P1065 study visit
* New diagnosis or suspected disease of the immune system since the last P1065 study visit
* Participant or legal guardian refuses further vaccine
* Participant requiring treatment with medications that were disallowed while on this study (see protocol)
* Grade 3 or higher toxicities (for example, Grade 3 seizure or allergic reaction) secondary to receipt of vaccine in previous version of P1065 meriting vaccine discontinuation, as determined by the IMPAACT P1065 Protocol Team and the site principal investigator
* Current immunomodulatory therapy, including IL-2, any interferon product, GM-CSF, or thalidomide [Note: G-CSF and erythropoietin are allowed]
* Current immunosuppressive therapy, including the equivalent of greater than or equal to 1 mg/kg/per day of prednisone in the 2 weeks preceding study entry
* Participants for whom long-term corticosteroid therapy (greater than or equal to 2 weeks) was anticipated were excluded [Note: non-steroidal anti-inflammatory agents and inhaled, intranasal and topical corticosteroids were allowed]
* A severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that required medical intervention, occurring within 24 hours of the first vaccine and potentially attributable to that first vaccine
* New diagnosis of any coagulation disorder that would contraindicate IM injections since the last P1065 study visit
* Breastfeeding
* Any new diseases which the investigators judged to be clinically significant (other than HIV infection) or clinically significant findings since enrollment into P1065 that, in the investigators' opinion, would have compromise the outcome of this study
* Any new greater than or equal to grade 3 clinical toxicity that is not related to vaccine and had not resolved within 2 weeks before entry into Step 3

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 384 (Actual)
Dates: Start 2007-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George K. Siberry, MD, MPH, Study Chair — Pediatric, Adolescent, and Maternal AIDS (PAMA) Branch, Eunice Kennedy Shriver National Institute of Child Health and Human Development, National Institutes of Health; Jorge Lujan-Zilbermann, MD, MS, Study Chair — Division of Infectious Diseases, Department of Pediatrics, University of South Florida College of Medicine
Locations (37):
- United States (35):
  - Usc La Nichd Crs, Alhambra, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - Children's Hospital of Los Angeles NICHD CRS, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - University of California, UC San Diego CRS, San Diego, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Harbor UCLA Medical Ctr. NICHD CRS, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Tulane Univ. New Orleans NICHD CRS, New Orleans, Louisiana
  - Univ. of Maryland Baltimore NICHD CRS, Baltimore, Maryland
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - Bronx-Lebanon CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Texas Children's Hospital CRS, Houston, Texas
  - Seattle Children's Research Institute CRS, Seattle, Washington
- Puerto Rico (2):
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Campos-Outcalt D. Meningococcal vaccine: New product, new recommendations. J Fam Pract. 2005 Apr;54(4):324-6. PMID 15833222
- [Background] Centers for Disease Control and Prevention (CDC). Update: Guillain-Barre syndrome among recipients of Menactra meningococcal conjugate vaccine--United States, June 2005-September 2006. MMWR Morb Mortal Wkly Rep. 2006 Oct 20;55(41):1120-4. PMID 17060898
- [Background] Keyserling H, Papa T, Koranyi K, Ryall R, Bassily E, Bybel MJ, Sullivan K, Gilmet G, Reinhardt A. Safety, immunogenicity, and immune memory of a novel meningococcal (groups A, C, Y, and W-135) polysaccharide diphtheria toxoid conjugate vaccine (MCV-4) in healthy adolescents. Arch Pediatr Adolesc Med. 2005 Oct;159(10):907-13. doi: 10.1001/archpedi.159.10.907. PMID 16203934
- [Background] Mehlhorn AJ, Balcer HE, Sucher BJ. Update on prevention of meningococcal disease: focus on tetravalent meningococcal conjugate vaccine. Ann Pharmacother. 2006 Apr;40(4):666-73. doi: 10.1345/aph.1G486. Epub 2006 Mar 7. PMID 16595570
- [Background] Platonov AE, Vershinina IV, Kuijper EJ, Borrow R, Kayhty H. Long term effects of vaccination of patients deficient in a late complement component with a tetravalent meningococcal polysaccharide vaccine. Vaccine. 2003 Oct 1;21(27-30):4437-47. doi: 10.1016/s0264-410x(03)00440-7. PMID 14505927
- [Background] Pearson IC, Baker R, Sullivan AK, Nelson MR, Gazzard BG. Meningococcal infection in patients with the human immunodeficiency virus and acquired immunodeficiency syndrome. Int J STD AIDS. 2001 Jun;12(6):410-1. doi: 10.1258/0956462011923237. PMID 11368827
- [Result] Siberry GK, Williams PL, Lujan-Zilbermann J, Warshaw MG, Spector SA, Decker MD, Heckman BE, Demske EF, Read JS, Jean-Philippe P, Kabat W, Nachman S; IMPAACT P1065 Protocol Team. Phase I/II, open-label trial of safety and immunogenicity of meningococcal (groups A, C, Y, and W-135) polysaccharide diphtheria toxoid conjugate vaccine in human immunodeficiency virus-infected adolescents. Pediatr Infect Dis J. 2010 May;29(5):391-6. doi: 10.1097/INF.0b013e3181c38f3b. PMID 20431379
- [Result] Spector SA, Qin M, Lujan-Zilbermann J, Singh KK, Warshaw MG, Williams PL, Jean-Philippe P, Fenton T, Siberry GK; IMPAACT P1065 Protocol Team. Genetic variants in toll-like receptor 2 (TLR2), TLR4, TLR9, and FCgamma receptor II are associated with antibody response to quadrivalent meningococcal conjugate vaccine in HIV-infected youth. Clin Vaccine Immunol. 2013 Jun;20(6):900-6. doi: 10.1128/CVI.00042-13. Epub 2013 Apr 17. PMID 23595505
- [Result] Lujan-Zilbermann J, Warshaw MG, Williams PL, Spector SA, Decker MD, Abzug MJ, Heckman B, Manzella A, Kabat B, Jean-Philippe P, Nachman S, Siberry GK; International Maternal Pediatric Adolescent AIDS Clinical Trials Group P1065 Protocol Team. Immunogenicity and safety of 1 vs 2 doses of quadrivalent meningococcal conjugate vaccine in youth infected with human immunodeficiency virus. J Pediatr. 2012 Oct;161(4):676-81.e2. doi: 10.1016/j.jpeds.2012.04.005. Epub 2012 May 22. PMID 22622049
- [Result] Siberry GK, Warshaw MG, Williams PL, Spector SA, Decker MD, Jean-Philippe P, Yogev R, Heckman BE, Manzella A, Roa J, Nachman S, Lujan-Zilbermann J; IMPAACT P1065 Protocol Team. Safety and immunogenicity of quadrivalent meningococcal conjugate vaccine in 2- to 10-year-old human immunodeficiency virus-infected children. Pediatr Infect Dis J. 2012 Jan;31(1):47-52. doi: 10.1097/INF.0b013e318236c67b. PMID 21987006

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: CD4%≥15, Age ≤11 to <25: Participants ≤11 to <25 years of age with CD4% at screening ≥15%; All receiving Quadrivalent meningococcal conjugate vaccine at entry, those who were eligible/randomized receiving Quadrivalent meningococcal conjugate vaccine at week 24, and 3 years.
  Quadrivalent meningococcal conjugate vaccine: MCV4 vaccine (4 µg each of meningococcal A, C, Y, and W-135 polysaccharides conjugated to approximately 48 µg of diphtheria toxoid protein carrier ) was given by injection intramuscularly at least once and no more than two times for each participant, depending on adverse reactions.
- Group 2: CD4%<15, Age ≤11 to <25: Participants ≤11 to <25 years of age with CD4% at screening <15%; All receiving Quadrivalent meningococcal conjugate vaccine at entry, those who were eligible receiving Quadrivalent meningococcal conjugate vaccine at week 24.
  Quadrivalent meningococcal conjugate vaccine: MCV4 vaccine (4 µg each of meningococcal A, C, Y, and W-135 polysaccharides conjugated to approximately 48 µg of diphtheria toxoid protein carrier ) was given by injection intramuscularly at least once and no more than two times for each participant, depending on adverse reactions.
- Group 3: Age ≥2 to <11, CD4%≥25: Participants ≥2 to <11 years of age with CD4% at screening ≥ 25%; All receiving Quadrivalent meningococcal conjugate vaccine at entry, those who were eligible receiving Quadrivalent meningococcal conjugate vaccine at week 24, and 3 years.
  Quadrivalent meningococcal conjugate vaccine: MCV4 vaccine (4 µg each of meningococcal A, C, Y, and W-135 polysaccharides conjugated to approximately 48 µg of diphtheria toxoid protein carrier ) was given by injection intramuscularly at least once and no more than two times for each participant, depending on adverse reactions.
Period: Steps 1 & 2
Arm/Group | Group 1: CD4%≥15, Age ≤11 to <25 | Group 2: CD4%<15, Age ≤11 to <25 | Group 3: Age ≥2 to <11, CD4%≥25
Started | 280 | 39 | 59
Completed | 259 | 32 | 57
Not Completed | 21 | 7 | 2
Not completed — Other eligibility failure | 1 | 1 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Not able to get to clinic | 7 | 4 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 0
Not completed — Not willing to adhere to regulations | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 2
Period: Step 3
Arm/Group | Group 1: CD4%≥15, Age ≤11 to <25 | Group 2: CD4%<15, Age ≤11 to <25 | Group 3: Age ≥2 to <11, CD4%≥25
Started | 152 (Not all participants from Steps 1/2 were eligible for Step 3) | 0 (Group 2 participants were not eligible for Step 3) | 40 (Not all participants from Steps 1/2 were eligible for Step 3)
Completed | 149 | 0 | 39
Not Completed | 3 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who started study treatment.
Groups:
- Group 1 (15<CD4%<25): Participants ≥11 to <25 years with 15<CD4%<25
- Group 1 (CD4%≥25): Participants ≥11 to <25 years with CD4%≥25
- Group 2: Participants ≥11 to <25 years with CD4%<15
- Group 3: Participants ≥ 2 to <11 years with CD4% ≥25
- Total: Total of all reporting groups
Arm/Group | Group 1 (15<CD4%<25) | Group 1 (CD4%≥25) | Group 2 | Group 3 | Total
Number analyzed (Participants) | 127 | 153 | 39 | 59 | 378
Age, Continuous [Median (Full Range); unit: years] | 18 [11 to 24] | 16 [11 to 24] | 20 [14 to 24] | 6 [2 to 10] | 16 [2 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 70 | 16 | 31 | 161
  Male | 83 | 83 | 23 | 28 | 217
Race [Number; unit: participants]
  Asian | 1 | 1 | 0 | 2 | 4
  Native Hawaiian or other Pacific islander | 1 | 0 | 0 | 1 | 2
  Black or African American | 72 | 69 | 22 | 34 | 197
  White | 47 | 75 | 14 | 21 | 157
  American Indian | 2 | 3 | 0 | 0 | 5
  More than One race | 0 | 3 | 2 | 0 | 5
  Unknown | 4 | 2 | 1 | 1 | 8
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 44 | 61 | 16 | 18 | 139
  Not Hispanic or Latino | 83 | 89 | 23 | 40 | 235
  Unknown | 0 | 3 | 0 | 1 | 4
Screening CD4% [Median (Full Range); unit: percent] | 20.0 [14.0 to 24.9] | 33.0 [25.0 to 53.1] | 8.5 [1.0 to 14.0] | 36.0 [25.0 to 56.0] | 27.9 [1.0 to 56.0]
Entry plasma HIV RNA viral load, copies/mL [Number; unit: participants]
  <400 copies/mL | 35 | 83 | 3 | 43 | 164
  ≥ 400 copies/mL | 92 | 70 | 36 | 16 | 214
CDC Classification at Study Entry [Number; unit: participants]
  C | 28 | 37 | 11 | 8 | 84
  Not C | 99 | 116 | 28 | 51 | 294
Antiretroviral (ARV) Treatment at Entry [Number; unit: participants]
  HAART with PI | 70 | 81 | 22 | 38 | 211
  HAART with NNRTI (no PI) | 14 | 34 | 3 | 14 | 65
  Other ARV | 6 | 8 | 1 | 1 | 16
  No ARV | 37 | 30 | 13 | 6 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Immunogenic Responders, With Response Defined as a 4-fold or Greater Increase in Serum Bactericidal Antibody Titers From Study Entry to Week 28 After 2 Doses of MCV-4.
Description: Serum bactericidal antibody titers were measured at study entry and Week 28 for each of the four serogroups in the MCV-4 vaccine. Response was defined as a 4-fold or greater increase from entry at Week 28.
Time Frame: Study entry and Week 28
Population: This outcome only includes participants who received 2 doses and had antibody data from both entry and Week 28.The number of participants analyzed for Group 1 (15<CD4%<25), Group 1 (CD4%≥25), Group 2, Group 3 are respectively:
  serogroup A: 49, 63, 20, 49 serogroup C: 47, 65, 18, 49 serogroup W-135: 47, 66, 19, 49 serogroup Y: 49, 66, 19, 49
Measure: Number; unit: participants
Groups:
- Group 1 (15<CD4%<25): Participants ≥11 to <25 years with 15<CD4%≤25
Arm/Group | Group 1 (15<CD4%<25) | Group 1 (CD4%≥25) | Group 2 | Group 3
Number analyzed (Participants) | 49 | 66 | 20 | 49
participants
  Week 28 reponders, serogroup A | 27 [0.87 to 0.99] | 60 [0.40 to 0.69] | 8 [0.19 to 0.64] | 43 [0.75 to 0.95]
  Week 28 reponders, serogroup C | 28 [0.44 to 0.74] | 49 [0.63 to 0.85] | 1 [0.001 to 0.27] | 39 [0.66 to 0.90]
  Week 28 reponders, serogroup W-135 | 36 [0.50 to 0.78] | 61 [0.70 to 0.90] | 0 [0 to 0.18] | 49 [0.93 to 1.00]
  Week 28 reponders, serogroup Y | 32 [0.62 to 0.88] | 54 [0.83 to 0.97] | 1 [0.001 to 0.25] | 41 [0.70 to 0.93]

2. Primary Outcome: Number of Participants With Short-term Immunogenicity, Defined as Number of Seroconverters at Week 4 (Those With at Least a 4-fold Rise in Meningococcal Serum Bactericidal Titers From Baseline)
Description: Serum bactericidal antibody titers were measured at study entry and Week 4 for each of the four serogroups in the MCV-4 vaccine. Response (seroconversion) was defined as a 4-fold or greater increase from entry at Week 4.
Time Frame: At Study entry, Week 4
Population: This outcome only includes participants who had antibody data from both entry and Week 4.The number of participants analyzed for Group 1 (15<CD4%<25), Group 1 (CD4%≥25), Group 2, Group 3 respectively are:
  serogroup A are 93, 129, 20, 49 serogroup C are 90, 130, 18, 49 serogroup W-135 are 91, 131, 19, 49 serogroup Y are 93, 131, 20, 49
Measure: Number; unit: participants
Groups:
- Group 3: Participants ≥ 2 to <11 years with CD4%≥25
Arm/Group | Group 1 (15<CD4%<25) | Group 1 (CD4%≥25) | Group 2 | Group 3
Number analyzed (Participants) | 93 | 131 | 20 | 49
participants
  Week 4 Seroconverters, serogroup A | 61 | 107 | 5 | 45
  Week 4 Seroconverters, serogroup C | 44 | 89 | 3 | 21
  Week 4 Seroconverters, serogroup W-135 | 66 | 118 | 6 | 48
  Week 4 Seroconverters, serogroup Y | 49 | 100 | 8 | 37

3. Primary Outcome: Long-term Immunogenicity, as Assessed by Number of Participants With Protective Levels of Antibody at Week 72
Description: Protective levels of antibody are titers ≥1:128.
Time Frame: Week 72
Population: Participants with antibody data at Week 72. The number of Participants analyzed for Group 1 (15<CD4%<25), Group 1 (CD4%≥25), Group 2, Group 3 respectively are:
  serogroup A are 82, 108, 18, 44 serogroup C are 78, 110, 16, 44 serogroup W-135 are 80, 110, 17, 44 serogroup Y are 82, 110, 18, 44
Measure: Number; unit: participants
Arm/Group | Group 1 (15<CD4%<25) | Group 1 (CD4%≥25) | Group 2 | Group 3
Number analyzed (Participants) | 82 | 110 | 18 | 44
participants
  Week 72 Responders, serogroup A | 39 | 82 | 4 | 35
  Week 72 Responders, serogroup C | 17 | 36 | 1 | 20
  Week 72 Responders, serogroup W-135 | 36 | 83 | 6 | 42
  Week 72 Responders, serogroup Y | 49 | 80 | 5 | 40

4. Primary Outcome: Number of Participants With Grade 3 or Higher Adverse Events Within 42 Days Following Dose 1 of the Vaccine.
Description: Adverse events were graded by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, dated December, 2004, Clarification August 2009, which is available on the RSC web site (http://rsc.tech-res.com/safetyandpharmacovigilance/). Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening, Grade 5 = death.
Time Frame: From administration of Dose 1 at week 0 to 42 days post-vaccination
Population: All participants who received Dose 1.
Measure: Number; unit: participants
Arm/Group | Group 1 (15<CD4%<25) | Group 1 (CD4%≥25) | Group 2 | Group 3
Number analyzed (Participants) | 127 | 153 | 39 | 59
participants | 3 | 1 | 3 | 0
Statistical Analysis 1: Comparison: Group 1 (15<CD4%<25) vs Group 1 (CD4%≥25) vs Group 2; The null hypothesis was that there would be no difference between CD4% strata; Test type: Superiority or Other; p = 0.03, Fisher Exact — Two-sided p-value <0.05 was specified as statistically significant a priori. There were no adjustments for multiple outcomes

5. Primary Outcome: Number of Participants With Reactions and Grade 3 or Higher Adverse Events Within 42 Days Following Dose 2 of the Vaccine.
Description: as for outcome 4
Time Frame: From administration of Dose 2 at week 24 to 6 weeks post-vaccination
Population: All participants who entered Step 2
Measure: Number; unit: participants
Arm/Group | Group 1 (15<CD4%<25) | Group 1 (CD4%≥25) | Group 2 | Group 3
Number analyzed (Participants) | 111 | 144 | 31 | 58
participants | 0 | 0 | 2 | 0
Statistical Analysis 1: Comparison: Group 1 (15<CD4%<25) vs Group 1 (CD4%≥25) vs Group 2; The null hypothesis was that there were no differences between CD4% strata; Test type: Superiority or Other; p = 0.01, Fisher Exact — Two sided-p-value <0.05 was specified as statistically significant a priori. No adjustment for multiple primary outcomes was made

6. Primary Outcome: Number of Participants With Immunogenicity at Step 3 Entry
Description: Immunogenicity was assessed for each serogroup by the number of participants with protective antibody levels (titers greater than or equal to 1:128)
Time Frame: At 3.5 years (Step 3 entry)
Population: All participants who had antibody data for Step 3 Week 0
Measure: Number; unit: participants
Groups:
- Group 1A: Participants ≥11 to <25 years with CD4%>15, 1 dose MCV4 vaccine
- Group 1B: Participants ≥11 to <25 years with CD4%>15, 2 doses MCV4 vaccine
Arm/Group | Group 1A | Group 1B | Group 3
Number analyzed (Participants) | 73 | 77 | 39
participants
  Immunogenicity, Serogroup A | 47 [.52 to .75] | 48 [.51 to .73] | 34 [.73 to .96]
  Immunogenicity, Serogroup C | 19 [.16 to .38] | 20 [.17 to .37] | 9 [.11 to .39]
  Immunogenicity, Serogroup W-135 | 30 [.30 to .53] | 35 [.34 to .57] | 23 [.42 to .74]
  Immunogenicity, Serogroup Y | 39 [.41 to .65] | 33 [.32 to .55] | 24 [.45 to .77]

7. Primary Outcome: Number of Participants With 4-fold Memory Response in Step 3
Description: Defined for each serogroup as a four-fold rise in antibody titers between booster dose (week 0) and week 1.
Time Frame: Step 3 entry and Week 1 post-booster vaccine
Population: Because response is a combination of memory and primary response, only participants with data for weeks 0, 1 and 4 are included.
Measure: Number; unit: participants
Arm/Group | Group 1A | Group 1B | Group 3
Number analyzed (Participants) | 73 | 65 | 36
participants
  4-fold memory responders, serogroup A | 54 [0.62 to 0.84] | 49 [0.61 to 0.83] | 33 [0.78 to 1.00]
  4-fold memory responders, serogroup C | 56 [0.65 to 0.86] | 50 [0.63 to 0.84] | 34 [0.81 to 0.99]
  4-fold memory responders, serogroup W-135 | 63 [0.76 to 0.93] | 55 [0.73 to 0.92] | 33 [0.78 to 0.98]
  4-fold memory responders, serogroup Y | 54 [0.62 to 0.84] | 51 [0.67 to 0.88] | 33 [0.78 to 0.98]

8. Primary Outcome: Number of Participants With Seropositive Memory Response (in Step 3)
Description: Seropositive memory response was defined for each serogroup by having protective antibody levels (titer >= 1:128) on Day 0 or change from seronegative to seropositive between booster dose (Day 0) and Day 7.
Time Frame: Step 3 entry and Week 1 post-booster vaccine
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Group 1A | Group 1B | Group 3
Number analyzed (Participants) | 73 | 65 | 36
participants
  Seropositive memory responder, serogroup A | 65 [0.80 to 0.95] | 61 [0.83 to 0.98] | 35 [0.85 to 1.00]
  Seropositive memory responder, serogroup C | 62 [0.75 to 0.92] | 55 [0.71 to 0.90] | 34 [0.81 to 0.99]
  Seropositive memory responder, serogroup W-135 | 65 [0.80 to 0.95] | 60 [0.80 to 0.96] | 34 [0.81 to 0.99]
  Seropositive memory responder, serogroup Y | 67 [0.83 to 0.97] | 57 [0.74 to 0.93] | 33 [0.78 to 0.98]

9. Primary Outcome: Number of Participants With Primary Response (in Step 3)
Description: Primary response was defined for each serogroup as a four-fold rise in Ab concentration between day 0 and day 28, but not between day 0 and day 7; OR a change from seronegative on day 0 to seropositive on day 28, but not between day 0 and day 7. Note: a primary response can only occur in the absence of any memory response.
Time Frame: Step 3 entry and Week 4 post-booster vaccine
Population: as for outcome 7
Measure: Number; unit: participants
Groups:
- Group 1B: Participants aged 11 to 24 with a CD4 percentage of or greater than 15%, 2 doses MCV4 vaccine
Arm/Group | Group 1A | Group 1B | Group 3
Number analyzed (Participants) | 73 | 65 | 36
participants
  Primary responder, serogroup A | 2 [0 to 0.10] | 2 [0 to 0.10] | 0 [0 to 0.10]
  Primary responder, serogroup C | 1 [0 to 0.07] | 1 [0 to 0.08] | 1 [0 to 0.15]
  Primary responder, serogroup W-135 | 1 [0 to 0.07] | 0 [0 to 0.05] | 2 [0.01 to 0.19]
  Primary responder, serogroup Y | 1 [0 to 0.07] | 2 [0 to 0.11] | 2 [0.01 to 0.19]

10. Secondary Outcome: Immunogenic Response to Serogroup C in Group 2
Description: Immunogenic response as assessed by number of participants with protective antibody titers (>= 1:128) to serogroup C in Group 2 (entry CD4%<15)
Time Frame: At Weeks 4, 28, and 72
Population: Group 2 participants with response data for weeks 4, 28 and 72
Measure: Number; unit: participants
Groups:
- Week 4: Group 2 participants at Week 4
- Week 28: Group 2 participants at Week 28 (4 weeks after second vaccination)
- Week 72: Group 2 participants at Week 72
Arm/Group | Week 4 | Week 28 | Week 72
Number analyzed (Participants) | 18 | 18 | 16
participants | 4 | 4 | 1

11. Secondary Outcome: Number of Participants With Protective Antibody Titers for Serogroup C at Step 3 Entry
Description: Number of participants with protective antibody titers (rSBA>=1:128) for serogroup C by treatment arm (1 vs. 2 doses) of Group 1 (entry CD4% >= 15) at Step 3 entry
Time Frame: At 3.5 years
Population: Group 1 and 3 participants at entry to Step 3
Measure: Number; unit: participants
Groups:
- Group 3: Age 2-<6: Participants 2 to <6 years with CD4%>=25
- Group 3: Age 6-<11: Participants 6 to <11 years with CD4%>=25
Arm/Group | Group 1A | Group 1B | Group 3: Age 2-<6 | Group 3: Age 6-<11
Number analyzed (Participants) | 73 | 65 | 20 | 16
participants | 19 | 17 | 3 | 6

12. Secondary Outcome: Immunologic Memory for Serogroup C by Treatment Arm (1 vs. 2 Doses)
Description: Evidence of immunologic memory according to each of the following definitions:
  1. Secondary (anamnestic) response defined as a four-fold rise in Ab titers between day 0 (booster dose) and day 7; or
  2. Seroprotection on day 0 or change from titer <1:128 to titer ≥1:128 (seroprotection) between day 0 and day 7.
Time Frame: At Week 1 post-booster vaccination
Population: Participants in Group 1 who entered Step 3
Measure: Number; unit: participants
Arm/Group | Group 1A | Group 1B
Number analyzed (Participants) | 73 | 65
participants | 65 | 61

13. Secondary Outcome: Immunologic Memory or Primary Response for Serogroup C by Treatment Arm
Description: Immunologic Memory defined as:
  1. Secondary (anamnestic) response defined as a four-fold rise in Ab titers between day 0 (booster dose) and day 7; or
  2. Seroprotection on day 0 or change from titer <1:128 to titer ≥1:128 (seroprotection) between day 0 and day 7.
  Primary Response defined as:
  1. A four-fold rise in Ab concentration between day 0 and day 28, but not between day 0 and day 7; or
  2. A change from titer <1:128 on day 0 to titer ≥1:128on day 28, but not between day 0 and day 7.
Time Frame: At Week 4 post-booster vaccination
Population: Group 1 participants who entered Step 3
Measure: Number; unit: participants
Arm/Group | Group 1A | Group 1B
Number analyzed (Participants) | 73 | 65
participants | 64 | 57

14. Secondary Outcome: Safety, as Assessed by Number of Participants With Reactions and Grade 3 or Higher Adverse Events Within 42 Days Following Step 3 Dose of the Vaccine.
Description: as for outcome 4
Time Frame: From administration of vaccination at Step 3 entry through 6 weeks post-vaccination
Population: All participants who were vaccinated at Step 3 entry
Measure: Number; unit: participants
Groups:
- Group 1: Participants ≤11 to <25 years of age with CD4% at screening ≥15%
- Group 3: Participants >=2 to <11 years of age with CD4% at screening ≥ 25%
Arm/Group | Group 1 | Group 3
Number analyzed (Participants) | 152 | 40
participants | 2 | 0

15. Primary Outcome: Number of Participants With Immunogenicity at Step 3 Weeks 4 and 24
Description: Immunogenicity was assessed by the number of participants with protective levels of antibody (titers greater than or equal to 1:128)
Time Frame: At Step 3 Weeks 4 and 24 post-booster vaccine
Population: Participants with data for Step 3 weeks 4 and 24. The numbers for Group 1 (1-dose), Group 1 (2-dose), and Group 3 respectively are:
  Week 4: 73, 71, 37 Week 24: 73, 70, 33
Measure: Number; unit: participants
Groups:
- Group 3: Participants ≥ 2 to <11 years with CD4% ≥25, 2 doses MCV4 vaccine
Arm/Group | Group 1A | Group 1B | Group 3
Number analyzed (Participants) | 73 | 79 | 38
participants
  Week 4 immunogenicity, serogroup A | 66 [0.81 to 0.96] | 67 [0.86 to 0.98] | 37 [0.86 to 1.00]
  Week 4 immunogenicity, serogroup C | 61 [0.73 to 0.91] | 60 [0.77 to 0.94] | 35 [0.78 to 0.98]
  Week 4 immunogenicity, serogroup W-135 | 67 [0.83 to 0.97] | 64 [0.82 to 0.97] | 37 [0.86 to 1.00]
  Week 4 immunogenicity, serogroup Y | 67 [0.83 to 0.97] | 62 [0.78 to 0.95] | 35 [0.78 to 0.98]
  Week 24 immunogenicity, serogroup A | 58 [0.70 to 0.89] | 59 [0.73 to 0.92] | 30 [0.75 to 0.98]
  Week 24 immunogenicity, serogroup C | 41 [0.44 to 0.68] | 46 [0.52 to 0.76] | 24 [0.53 to 0.86]
  Week 24 immunogenicity, serogroup W-135 | 57 [0.67 to 0.87] | 53 [0.63 to 0.85] | 32 [0.84 to 1.00]
  Week 24 immunogenicity, serogroup Y | 58 [0.68 to 0.88] | 52 [0.61 to 0.84] | 31 [0.79 to 0.99]

ADVERSE EVENTS:
Time Frame: From study entry through Step 3, week 24 (4 years )
Description: All vaccine-related Grade ≥ 3 toxicities, and any new Grade 2 or higher neuromuscular weakness occurring within 42 days of vaccination were reported. Adverse events were graded by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, dated December, 2004, Clarification August 2009.
Groups:
- Group 1 (15<CD4%≤25): Participants ≥11 to <25 years with 15<CD4%≤25
Arm/Group | Group 1 (15<CD4%≤25) | Group 1 (CD4%≥25) | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 4/127 | 5/153 | 5/39 | 2/59
Other Adverse Events (participants affected / at risk) | 94/127 | 113/153 | 33/39 | 47/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (15<CD4%≤25) (N=127) | Group 1 (CD4%≥25) (N=153) | Group 2 (N=39) | Group 3 (N=59)
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (15<CD4%≤25) (N=127) | Group 1 (CD4%≥25) (N=153) | Group 2 (N=39) | Group 3 (N=59)
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 10 | 7 | 2 | 4
Conjunctivitis (Eye disorders) | 3 | 3 | 3 | 3
Eye discharge (Eye disorders) | 0 | 1 | 2 | 1
Eye pain (Eye disorders) | 0 | 2 | 3 | 0
Ocular hyperaemia (Eye disorders) | 0 | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 11 | 14 | 7 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 4 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 4 | 3
Nausea (Gastrointestinal disorders) | 7 | 7 | 2 | 2
Oral pain (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 7 | 9 | 4 | 4
Adverse event (General disorders) | 14 | 12 | 0 | 8
Chest pain (General disorders) | 7 | 4 | 3 | 1
Oedema peripheral (General disorders) | 1 | 1 | 3 | 0
Pyrexia (General disorders) | 13 | 11 | 6 | 12
Acute sinusitis (Infections and infestations) | 9 | 6 | 2 | 2
Bronchitis (Infections and infestations) | 3 | 4 | 2 | 4
Escherichia urinary tract infection (Infections and infestations) | 0 | 3 | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 3
Herpes zoster (Infections and infestations) | 11 | 3 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 0 | 3
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 3 | 0
Oral candidiasis (Infections and infestations) | 3 | 1 | 7 | 0
Otitis externa (Infections and infestations) | 3 | 1 | 2 | 1
Otitis media acute (Infections and infestations) | 7 | 8 | 3 | 5
Pharyngitis (Infections and infestations) | 5 | 8 | 4 | 4
Pneumonia (Infections and infestations) | 5 | 4 | 5 | 3
Subcutaneous abscess (Infections and infestations) | 3 | 0 | 3 | 0
Tinea capitis (Infections and infestations) | 0 | 2 | 1 | 3
Vulvovaginitis trichomonal (Infections and infestations) | 2 | 0 | 2 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 6 | 4 | 6 | 0
Neutrophil count decreased (Investigations) | 31 | 36 | 12 | 19
Platelet count decreased (Investigations) | 6 | 5 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 8 | 4 | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 5 | 1 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 5 | 0
Headache (Nervous system disorders) | 14 | 13 | 3 | 5
Syncope (Nervous system disorders) | 0 | 1 | 2 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 6 | 10 | 2 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 3 | 0 | 0 | 9
Major depression (Psychiatric disorders) | 4 | 3 | 5 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 7 | 6 | 3 | 0
Vaginal discharge (Reproductive system and breast disorders) | 9 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 23 | 3 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 1 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 13 | 7 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 1 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1 | 5
Acne (Skin and subcutaneous tissue disorders) | 12 | 10 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 7 | 4 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights